CLINICAL TRIAL: NCT02784496
Title: Open-Label Roll-Over Study to Assess the Long-Term Safety and Efficacy of Ruxolitinib in Subjects With Myelofibrosis
Brief Title: Long-Term Side Effects of Ruxolitinib in Treating Patients With Myelofibrosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2015-0872; NCI-2016-01181 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2015-0872 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2016-05-20; First posted 2016-05-27 (Estimated); Results first posted 2025-08-29 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2025-08

CONDITIONS: Myelofibrosis
MeSH Terms: conditions — Primary Myelofibrosis | interventions — ruxolitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (ruxolitinib, follow-up) (Experimental): Patients continue to receive ruxolitinib PO QD or BID. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients undergo follow-up assessment for safety over 10 minutes every 3 cycles.
  Interventions: Other: Long-term Follow-up; Other: Quality-of-Life Assessment; Drug: Ruxolitinib

INTERVENTIONS:
Other: Long-term Follow-up — Undergo follow-up assessment
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Drug: Ruxolitinib — Given PO
  Other Names: INCB-18424; INCB18424; Oral JAK Inhibitor INCB18424

SUMMARY:
This phase II trial studies the long-term side effects of ruxolitinib in treating patients with myelofibrosis. Collecting data about the long-term safety and tolerability of ruxolitinib may better help future patients with myelofibrosis.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To collect long term safety and tolerability data in patients with myelofibrosis previously treated with ruxolitinib on protocol 2007-0169.

OUTLINE:

Patients continue to receive ruxolitinib orally (PO) once daily (QD) or twice daily (BID). Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients undergo follow-up assessment for safety over 10 minutes every 3 cycles.

ELIGIBILITY:
Inclusion Criteria:

1. Currently enrolled in study 2007-0169 and benefiting from therapy as determined by treating physician
2. Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1, or 2 at enrollment of this study
3. Ability and agreement to attend protocol-specified visits at the study site
4. Able to comprehend and willing to sign the informed consent form
5. Negative pregnancy test in females of childbearing potential; male patients with female partners of child-bearing potential and female patients of childbearing potential are required to use two forms of acceptable contraception, including one barrier method, during their participation in the study and for 30 days following last dose; acceptable forms of contraception include 1 highly effective method such as an intrauterine device (IUD), hormonal (birth control pills, injections, or implants), tubal ligation, or partner's vasectomy and at least 1 additional approved barrier method such as a latex condom, diaphragm, or cervical cap; female patients of childbearing potential must not be breast-feeding or planning to breast feed and must have a negative pregnancy test 7 days before first study treatment

Exclusion Criteria:

1. none

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2016-09-29 (Actual); Primary Completion 2024-01-23 (Actual); Study Completion 2024-01-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Prithviraj Bose, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment (Ruxolitinib, Follow-up)
Started | 8
Completed | 8
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Ruxolitinib, Follow-up)
Number analyzed (Participants) | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 0
  >=65 years | 8
Age, Continuous [Median (Full Range); unit: years] | 73 [68 to 78]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 8
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 8

OUTCOME MEASURES:

1. Primary Outcome: Most Common Treatment Related Adverse Events
Description: A review of the most common adverse events related to study medication will be performed. Will follow standard reporting guidelines for adverse events. Safety data will be summarized by the number of participants affected.
Time Frame: to the date of failure or death from any cause, Up to 7 years, 3 months and 24 days
Measure: Number; unit: participants
Arm/Group | Treatment (Ruxolitinib, Follow-up)
Number analyzed (Participants) | 8
participants
  Infections | 1
  Headache | 1
  Fatigue | 2
  Dizziness | 1

ADVERSE EVENTS:
Time Frame: Up to the date of failure or death from any cause, up to 7 years, 3 months and 24 days.
Arm/Group | Treatment (Ruxolitinib, Follow-up)
All-Cause Mortality (participants affected / at risk) | 2/8
Serious Adverse Events (participants affected / at risk) | 6/8
Other Adverse Events (participants affected / at risk) | 8/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Ruxolitinib, Follow-up) (N=8)
Atrial fibrillation (Cardiac disorders) | 1 (2)
Fall (Injury, poisoning and procedural complications) | 1 (1)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Headache (General disorders) | 1 (1)
Hypertension (Vascular disorders) | 1 (1)
Intracranial hemorrhage (Nervous system disorders) | 1 (1)
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 (1)
Lung infection (Infections and infestations) | 2 (2)
Musculoskeletal and connective tissue disorder (Musculoskeletal and connective tissue disorders) | 2 (2)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (5)
Nervous system disorders (Nervous system disorders) | 1 (1)
Non-cardiac chest pain (General disorders) | 1 (1)
Renal calculi (Renal and urinary disorders) | 1 (1)
Sepsis (Infections and infestations) | 2 (3)
Skin infection (Infections and infestations) | 2 (2)
Surgical and medical procedures (Surgical and medical procedures) | 3 (3)
Urinary tract infection (Renal and urinary disorders) | 3 (4)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Ruxolitinib, Follow-up) (N=8)
Alanine aminotransferase increased (Investigations) | 2 (2)
Alkaline phosphatase increased (Investigations) | 1 (1)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Anorexia (Metabolism and nutrition disorders) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 (5)
Aspartate aminotransferase increased (Investigations) | 3 (4)
Atrial fibrillation (Cardiac disorders) | 1 (1)
Bloating (Gastrointestinal disorders) | 1 (1)
Bruising (Injury, poisoning and procedural complications) | 1 (1)
Chills (General disorders) | 1 (1)
Conjunctivitis (Infections and infestations) | 1 (1)
Constipation (Gastrointestinal disorders) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Creatinine increased (Investigations) | 2 (4)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Dizziness (Nervous system disorders) | 1 (3)
Dysarthria (Nervous system disorders) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Edema (General disorders) | 5 (6)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 2 (2)
Fatigue (General disorders) | 3 (3)
Fever (General disorders) | 1 (1)
Gait disturbance (General disorders) | 2 (2)
Gastrointestinal disorders (Gastrointestinal disorders) | 3 (4)
General disorders and administration site conditions (General disorders) | 1 (1)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 3 (4)
Hip fracture (Injury, poisoning and procedural complications) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1)
Hyperkalemia (Metabolism and nutrition disorders) | 2 (3)
Hypernatremia (Metabolism and nutrition disorders) | 1 (2)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (1)
Hypophosphatemia (Metabolism and nutrition disorders) | 1 (1)
Infection (Infections and infestations) | 2 (4)
Infections and infestations (Infections and infestations) | 1 (1)
Injury, poisoning and procedural complications (Injury, poisoning and procedural complications) | 3 (3)
Insomnia (Psychiatric disorders) | 1 (1)
Investigations (Investigations) | 5 (9)
Localized edema (General disorders) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2)
Myositis (Musculoskeletal and connective tissue disorders) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (2)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Night blindness (Eye disorders) | 1 (1)
Pain (General disorders) | 4 (9)
Paresthesia (Nervous system disorders) | 1 (1)
Peripheral motor neuropathy (Nervous system disorders) | 3 (3)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1)
Reproductive system and breast disorders (Reproductive system and breast disorders) | 1 (1)
Respiratory, thoracic and mediastinal disorders (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Skin and subcutaneous tissue disorders (Skin and subcutaneous tissue disorders) | 2 (6)
Surgical and medical procedures (Surgical and medical procedures) | 1 (1)
Urinary frequency (Renal and urinary disorders) | 1 (1)
Vascular disorders (Vascular disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-05-02): https://cdn.clinicaltrials.gov/large-docs/96/NCT02784496/Prot_SAP_000.pdf